CLINICAL TRIAL: NCT04955171
Title: Outcome of Brolucizumab-dbll and Aflibercept Intravitreal Injection in the Treatment of Diabetic Macular Edema
Brief Title: BEOVU Versus Eylea in the Treatment of Diabetic Macular Edema
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Associate Professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hamaky15
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Macular Edema
Keywords: BEOVU; Eylea; diabetic macular edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEOVU (Active Comparator): Intravitreal injection of BEOVU 3 loading injections( monthly) then under treat and extent regimen
  Interventions: Drug: BEOVU intravitreal injection
- Eylea (Active Comparator): Intravitreal injection of Eylea 3 loading injections( monthly) then under treat and extent regimen
  Interventions: Drug: BEOVU intravitreal injection

INTERVENTIONS:
Drug: BEOVU intravitreal injection — BEOVU intravitreal injection
  Other Names: Brolucizumab-Dbll intravitreal injection

SUMMARY:
Diabetic macular edema degeneration occur is a vision threatening condition. The investigators compare the efficacy of BEOVU and Eylea intravitreal treatment in the management

DETAILED DESCRIPTION:
Baseline ,and postoperative 1 ,6 and 12 months full ophthalmic examination was done. Procedure included randomized intravitreal injection of Brolucizumab(BEOVU®, Genentech, South Francisco, CA) and of aflibercept (Eylea;Regeneron, Tarrytown,NY)

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema

Exclusion Criteria:

* other causes of macular edema
* other macular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 12 months
  Change in BCVA in LOG MARS(logarithm minimum angle of resolution

CONTACTS AND LOCATIONS:
Overall Officials: TAREK ELHAMAKY, MD, Principal Investigator — Benha University
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
by direct contact through email
Supporting Information: Study Protocol, SAP
Time Frame: UNLIMITED